CLINICAL TRIAL: NCT07202481
Title: Effects of Chronic Ingestion of Fructooligosaccharide and Psyllium on Intestinal Transit Time in Women Diagnosed With Functional Constipation: A Randomized, Crossover, Double-Blind Clinical Trial
Brief Title: Chronic Ingestion of Fructooligosaccharide and Psyllium on Intestinal Transit in Women With Functional Constipation: A Randomized Crossover Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Max Nutri (Unknown)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 85835125.9.0000.5149
Record Dates: First submitted 2025-09-15; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Constipation - Functional
MeSH Terms: interventions — fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber A (Experimental): In this arm, participants start by undergoing scintigraphic imaging and data collection for the control period. Then, in a randomized order, they receive Fiber A for 6 days, at a dose of 20 g per day divided into two 10 g doses, after which scintigraphic imaging and data collection are repeated. Following a 7-day washout period, participants begin Fiber B consumption, also at 20 g per day divided into two 10 g doses, and return for new scintigraphic imaging and data collection.
  Interventions: Dietary Supplement: Psyllium powder
- Fiber B (Experimental): In this arm, participants start by undergoing scintigraphic imaging and data collection for the control period. Then, in a randomized order, they receive Fiber B for 6 days, at a dose of 20 g per day divided into two 10 g doses, after which scintigraphic imaging and data collection are repeated. Following a 7-day washout period, participants begin Fiber A consumption, also at 20 g per day divided into two 10 g doses, and return for new scintigraphic imaging and data collection.
  Interventions: Dietary Supplement: Fructooligosaccharide

INTERVENTIONS:
Dietary Supplement: Psyllium powder — Psyllium powder: soluble fiber gel forming, provided at 20 g per day (two doses of 10 g each)
  Arms: Fiber A
Dietary Supplement: Fructooligosaccharide — Fructooligosaccharide: prebiotic, provided at 20 g per day (two doses of 10 g each)
  Arms: Fiber B

SUMMARY:
The goal of this clinical trial is to evaluate the effect of dietary fibers in the treatment of functional constipation in women. It will also assess the potential side effects associated with fiber consumption. The main questions it aims to answer are:

* In women with constipation who do not consume adequate dietary fiber, does supplementation help improve bowel function?
* Among the fibers studied, is there any hierarchy of effect in the treatment of constipation (i.e., is one more effective than the other)?

The researchers will compare the effects of the two dietary fibers against each other and against a control to evaluate their impact.

Participants will:

* Consume 20 g of fiber daily for 6 days, divided into two doses of 10 g each.
* Attend a nuclear medicine visit at the end of each 6-day fiber period to perform scintigraphy.
* Keep a daily record of bowel habits and dietary intake.

ELIGIBILITY:
Inclusion Criteria

* Female participants aged 18-59 years.
* Willingness to sign the Informed Consent Form .
* No restrictions on the consumption of egg or gluten.
* No history or diagnosis of gastrointestinal diseases other than functional constipation.
* Non-smokers.
* No use of prebiotics, probiotics, synbiotics, or antibiotics at least 10 days prior to the study.
* No previous surgery affecting gastrointestinal transit.
* Willingness to discontinue the use of laxatives at least 4 days prior to scintigraphic imaging.
* Participants who do not consume adequate dietary fiber (25-30 g/day) as assessed by dietary recall.
* No confirmed or suspected pregnancy during the study.
* No self-reported menopause

Exclusion Criteria

* Diagnosis of diabetes, severe hyperthyroidism, or hypothyroidism.
* Use of opioid medications.
* Delayed gastric emptying at 4 hours during the placebo period (participants meeting this criterion will be excluded from final analysis).

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Colonic transit time | This outcome will be assessed at the end of the 6-day consumption period of the fibers of interest.
  Colonic transit time will be measured using scintigraphy 24 hours after ingestion of the radiolabeled test meal.

SECONDARY OUTCOMES:
Gastric emptying | This outcome will be assessed at the end of the 6-day consumption period of each fiber of interest
  Gastric emptying will be evaluated using scintigraphy, with images obtained immediately after ingestion of the radiolabeled test meal and then hourly for 6 hours.
Bowel function | The outcome will be assessed throughout the intervention period, during the 6-day consumption of the fibers of interest.
  Through questionnaires, the number of bowel movements and gastrointestinal symptoms experienced during the intervention period will be assessed
Quality of life assessment | Assessed at baseline and following each treatment phase of the crossover trial
  Using a validated questionnaire, the impact of constipation on the quality of life of women with constipation will be assessed.
Fecal microbiota | Baseline and at the end of each 6-day intervention period
  Fecal samples will be collected before and after the intervention to assess the gut microbiota and short-chain fatty acids.
Fecal Short chain fatty acids | Baseline and at the end of each 6-day intervention period
  Fecal samples will be collected before and after the intervention to assess the short-chain fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Simone de Vasconcelos Generoso, PhD, Principal Investigator — Department of Nutrition, Federal University of Minas Gerais
Locations (1):
- School of Nursing, Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No